CLINICAL TRIAL: NCT01074411
Title: A Phase I Pharmacokinetic Study of Intraperitoneal CTEP-Supplied Agent Bortezomib (PS-341, NSC 681239) and Carboplatin (NSC# 241240) in Patients With Persistent or Recurrent Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Brief Title: Intraperitoneal Bortezomib and Carboplatin in Treating Patients With Persistent or Recurrent Ovarian Epithelial Cancer, Fallopian Tube Cancer, or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02014; NCI-2011-02014 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000665312; GOG-9924 (Other: NRG Oncology); GOG-9924 (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2010-02-23; First posted 2010-02-24 (Estimated); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Fallopian Tube Clear Cell Adenocarcinoma; Fallopian Tube Endometrioid Adenocarcinoma; Fallopian Tube Mucinous Adenocarcinoma; Fallopian Tube Serous Adenocarcinoma; Fallopian Tube Transitional Cell Carcinoma; Ovarian Brenner Tumor; Ovarian Clear Cell Adenocarcinoma; Ovarian Clear Cell Cystadenocarcinoma; Ovarian Endometrioid Adenocarcinoma; Ovarian Mucinous Adenocarcinoma; Ovarian Mucinous Cystadenocarcinoma; Ovarian Seromucinous Carcinoma; Ovarian Serous Adenocarcinoma; Ovarian Serous Cystadenocarcinoma; Ovarian Transitional Cell Carcinoma; Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma; Undifferentiated Fallopian Tube Carcinoma; Undifferentiated Ovarian Carcinoma
MeSH Terms: conditions — Brenner Tumor; Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Bortezomib; Carboplatin

ARMS (1):
- Treatment (bortezomib, carboplatin) (Experimental): Patients receive bortezomib IP and carboplatin IP on day 1. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bortezomib; Drug: Carboplatin; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Drug: Bortezomib — Given IP
  Other Names: [(1R)-3-Methyl-1-[[(2S)-1-oxo-3-phenyl-2-[(pyrazinylcarbonyl)amino]propyl]amino]butyl]boronic Acid; LDP 341; MLN341; PS-341; PS341; Velcade
Drug: Carboplatin — Given IP
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of intraperitoneal bortezomib when given together with intraperitoneal carboplatin in treating patients with ovarian epithelial cancer, fallopian tube cancer, or primary peritoneal cancer that is persistent or has come back. Bortezomib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Bortezomib may help carboplatin work better by making tumor cells more sensitive to the drug. Infusing bortezomib and carboplatin directly into the abdomen (intraperitoneal) may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum-tolerated dose (MTD) and dose-limiting toxicities (DLTs) of intraperitoneal (IP) bortezomib (BTZ) when administered with intraperitoneal carboplatin in women with epithelial ovarian, fallopian tube, or primary peritoneal cancer that is persistent or recurrent and who have failed primary therapy and at least one second-line therapy.

II. To examine the safety of administering BTZ in combination with carboplatin by the IP route.

SECONDARY OBJECTIVES:

I. To estimate objective tumor response rate as determined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria.

II. To determine the pharmacokinetic profile of BTZ and carboplatin when administered intraperitoneally once every 21 days.

III. To characterize the frequency of carboplatin hypersensitivity reactions (HSR) when administered as an intraperitoneal infusion in the context of recurrent ovarian cancer.

OUTLINE: This is a dose-escalation study of bortezomib.

Patients receive bortezomib intraperitoneally (IP) and carboplatin IP on day 1. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have recurrent or persistent epithelial ovarian, fallopian tube, or primary peritoneal cancer; histologic documentation of the original primary tumor is required via the pathology report

  * Patients with the following histologic epithelial cell types are eligible: serous adenocarcinoma, endometrioid adenocarcinoma, mucinous adenocarcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial carcinoma, transitional cell carcinoma, malignant Brenner's tumor, or adenocarcinoma not otherwise specified (N.O.S)
* Patients must have either measurable disease or detectable disease:

  * Measurable disease will be defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1; measureable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest dimension to be recorded); each lesion must be >= 10 mm when measured by computed tomography (CT), magnetic resonance imaging (MRI) or caliper measurement by clinical exam; or >= 20 mm when measured by chest x-ray; lymph nodes must be >= 15 mm in short axis when measured by CT or MRI
  * Detectable disease is defined in a patient as one who does not have measurable disease but has at least one of the following conditions:

    * Baseline values of cancer antigen (CA)-125 at least twice the upper limit of normal
    * Ascites and/or pleural effusion attributed to tumor
    * Solid and/or cystic abnormalities on radiographic imaging that do not meet RECIST 1.1 definitions for target lesions
  * In addition, patients are allowed to undergo surgical cytoreduction of relapsed disease as proof of detectable disease at the discretion of their treating physician; if performed to allow participation in this protocol, the operative and pathology reports will be required for submission
* Patients must have a Gynecologic Oncology Group (GOG) performance status 0, 1, or 2
* Recovery from effects of recent surgery, radiotherapy, or chemotherapy

  * Patients should be free of active infection requiring antibiotics (with the exception of uncomplicated urinary tract infection [UTI])
  * Any hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to registration; continuation of hormone replacement therapy is permitted
  * Any other prior therapy directed at the malignant tumor, including biological and immunologic agents, must be discontinued at least three weeks prior to registration
* Patients must have had one prior platinum-based chemotherapeutic regimen for management of primary disease containing carboplatin, cisplatin, or another organoplatinum compound; this initial treatment may have included non-cytotoxic therapy, intraperitoneal therapy, consolidation, or extended therapy administered after surgical or non-surgical assessment

  * Patients are required to receive, one additional cytotoxic regimen for management of recurrent or persistent disease
  * Patients are allowed to receive, but are not required to receive, two additional cytotoxic regimens for management of recurrent or persistent disease (maximum number of prior cytotoxic regimens including primary therapy is 4); patients are allowed to receive, but are not required to receive, biologic (non-cytotoxic) therapy either alone or as part of the cytotoxic regimens for management of recurrent or persistent disease
* Absolute neutrophil count (ANC) greater than or equal to 1,500/mcl, equivalent to the National Cancer Institute (NCI) Common Terminology Criteria (CTCAE) version 4 grade 1
* Platelets greater than or equal to 100,000/mcl
* Creatinine less than or equal to institutional upper limit of normal (ULN)
* Bilirubin less than or equal to 1.5 x ULN (per the NCI CTCAE version 4 grade 1)
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) less than or equal to 3 x ULN (per the active version of the NCI CTCAE grade 1)
* Alkaline phosphatase less than or equal to 2.5 x ULN (per the NCI CTCAE version 4 grade 1)
* Neuropathy (sensory and motor) less than or equal to the NCI CTCAE version 4 grade 1
* Prothrombin time (PT) such that international normalized ratio (INR) is =< 1.5 x ULN (or an in-range INR, usually between 2 and 3, if a patient is on a stable dose of therapeutic warfarin)
* Partial thromboplastin time (PTT) =< 1.5 x ULN (heparin, low molecular weight heparin, or alternative anticoagulants are acceptable)
* Patients who have met the pre-entry requirements
* An approved informed consent and authorization permitting release of personal health information must be signed by the patient or guardian
* Patients of childbearing potential must have a negative serum pregnancy test prior to the study entry and be practicing an effective form of contraception
* Patients in this trial may receive ovarian estrogen +/- progestin replacement therapy as indicated at the lowest effective dose(s) for control of menopausal symptoms at any time, but not progestins for management of anorexia while on protocol directed therapy or prior to disease progression

Exclusion Criteria:

* Patients who have had prior therapy with bortezomib
* Patient with a history of other invasive malignancies, with the exceptions of non-melanoma skin cancer and localized breast cancer, are excluded if there is any evidence of other malignancy being present within the last five years; patients are also excluded if their previous cancer treatment contraindicates this protocol therapy
* Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis OTHER THAN for the treatment of ovarian cancer are excluded; prior radiation for localized cancer of the breast, head and neck, or skin is permitted, provided that it was completed more than three years prior to registration, and the patient remains free of recurrent or metastatic disease
* Patients who have received prior chemotherapy for any abdominal or pelvic tumor OTHER THAN for the treatment of ovarian cancer are excluded

  * Patients may have received prior adjuvant chemotherapy for localized breast cancer, provided that it was completed more than three years prior to registration, and that the patient remains free of recurrent or metastatic disease
* Patients with known brain metastases are excluded
* History of allergic reactions attributed to carboplatin or compounds of similar chemical or biologic composition to bortezomib including boron or mannitol
* Patients with synchronous primary endometrial cancer, or a past history of primary endometrial cancer, are excluded, unless all of the following conditions are met: stage not greater than I-B; no more than superficial myometrial invasion, without vascular or lymphatic invasion; no poorly differentiated subtypes, including papillary serous, clear cell or other International Federation of Gynecology and Obstetrics (FIGO) grade 3 lesions
* Patients with a history of prior myocardial infarction in the last 12 months or patients with new electrocardiographic evidence of acute ischemia or new conduction abnormalities are ineligible
* Uncontrolled concurrent illness including but not limited to ongoing or active infection that requires parenteral antibiotics, acute hepatitis, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients with insulin-dependent diabetes will be excluded
* Concomitant medications known to inhibit or induce cytochrome P450, family 3, subfamily A, polypeptide 4 (3A4) are to be avoided

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2010-04-05 (Actual); Primary Completion 2014-04-04 (Actual); Study Completion 2018-01-27 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicities defined by drug-related adverse events which occur in association with the first course of treatment as evaluated by the NCI CTCAE version 4 unless clearly unrelated to study drugs (e.g., disease progression) | 21 days
Frequency and severity of toxicities as assessed by NCI CTCAE version 4 | Up to 1 year

SECONDARY OUTCOMES:
Objective tumor response (complete and partial response) | Up to 1 year
  Objective tumor response will be tabulated by regimen.
Progression free survival | Time from study entry to time of progression or death, whichever occurs first, assessed up to 1 year
  Will be summarized using Kaplan-Meier plots.
Pharmacokinetic parameters | 10 minutes prior to infusion; immediately following infusion; 15, 30 and 60 minutes after infusion; immediately following carboplatin; 90 minutes after infusion; and 2, 4, and 6 hours after infusion
  Descriptive analysis will be given for the pharmacokinetic parameters of bortezomib and carboplatin.

CONTACTS AND LOCATIONS:
Overall Officials: Don Dizon, Principal Investigator — NRG Oncology
Locations (14):
- United States (14):
  - Hartford Hospital, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Washington University School of Medicine, St Louis, Missouri
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Women and Infants Hospital, Providence, Rhode Island
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia

REFERENCES:
- [Derived] Jandial DA, Brady WE, Howell SB, Lankes HA, Schilder RJ, Beumer JH, Christner SM, Strychor S, Powell MA, Hagemann AR, Moore KN, Walker JL, DiSilvestro PA, Duska LR, Fracasso PM, Dizon DS. A phase I pharmacokinetic study of intraperitoneal bortezomib and carboplatin in patients with persistent or recurrent ovarian cancer: An NRG Oncology/Gynecologic Oncology Group study. Gynecol Oncol. 2017 May;145(2):236-242. doi: 10.1016/j.ygyno.2017.03.013. Epub 2017 Mar 22. PMID 28341300